CLINICAL TRIAL: NCT02420106
Title: Effect of Osteopathic Manipulative Medicine on Motor Function and Quality of Life in Cervical Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BHS-983
Record Dates: First submitted 2014-02-18; First posted 2015-04-17 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Cervical Dystonia
Keywords: cervical dystonia; neck pain; OMM; spasmodic torticollis
MeSH Terms: conditions — Torticollis; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMM alone (Active Comparator): Subjects who are not receiving botulinum treatment consenting to Osteopathic Manipulative Medicine intervention
  Interventions: Procedure: Osteopathic Manipulative Medicine
- OMM plus Botulinum (Active Comparator): Subjects who are receiving botulinum treatment and will have osteopathic manipulative medicine intervention.
  Interventions: Procedure: Osteopathic Manipulative Medicine

INTERVENTIONS:
Procedure: Osteopathic Manipulative Medicine — Osteopathic manipulative medicine involves manual technique to joints and soft tissue to improve movement.

SUMMARY:
The purpose of the proposed research is to determine if Osteopathic manipulative medicine (OMM) used alone or in combination with the standard treatment of botulinum toxin intramuscular injections improves motor function and quality of life amongst people with cervical (neck) dystonia.

DETAILED DESCRIPTION:
Cervical dystonia, also called spasmodic torticollis, is a type of neurological disorder characterized by spastic muscles in the neck that is largely underdiagnosed despite its progression to disability during midlife. Cervical dystonia occurs in at least 0.390% of the United States population in 2007 (390 per 100,000). Symptoms commonly include stiffness, pain, headaches, difficulty swallowing, fatigue, and difficulty walking. The current standard treatment is intramuscular botulinum toxin injection every 90 days. The effect of the botulinum toxin increases gradually, and then it decreases until there is little to no effect at 90 days post-injection. The purpose of the proposed research is to determine if Osteopathic manipulative medicine (OMM) used in combination with the standard treatment of botulinum toxin intramuscular injections improves motor function and quality of life amongst people with cervical dystonia.

The investigators propose to use Vicon 3-dimensional gait and posture analysis to determine the biomechanics of subjects with primary cervical dystonia to compare with full body complaints from a standard spasmodic torticollis/cervical dystonia questionnaire as well as the osteopathic structural exam. These measures will be assessed before and after four OMM treatments. In addition, the investigators propose to use osteopathic manual medicine along with botulinum toxin injection to improve the subjects' pain and motor function as evaluated by Vicon 3-dimensional gait and posture analysis and questionnaire regarding quality of life. Preliminary case reports suggest that Osteopathic manipulative medicine without botulinum toxin injections improved pain, posture, gait, and quality of life in four adult subjects as well as improved head tilt in two children (two- and five-years old). The central hypothesis is that osteopathic manual medicine will significantly improve the range of motion, motor function, and quality of life of subjects with primary cervical dystonia.

Aims:

Aim I. To determine 3-Dimensional gait and posture biomechanics of subjects with untreated primary cervical dystonia while walking, and to investigate the effectiveness of OMM in treating abnormal biomechanics in these subjects.

Hypothesis I: People with cervical dystonia have similar abnormalities in posture and structural exam that significantly alters their gait and full body motor function that can be significantly improved with OMM.

Experimental approach: Motor function will be assessed by Vicon 3-Dimensional analysis using 34 of the subjects while walking will depict stride length and arm swing on each side of the body as well as the posture of the shoulder and pelvic girdle with reference to the coronal, transverse, and sagittal planes. Quality of life will be assessed by the Cervical Dystonia Impact Profile (CDIP)-58 questionaire. Four weekly OMM diagnosis and treatment will be done, and then, motor function and quality of life will be reassessed. Total participation in the study is expected to last for 5-7 weeks.

Expected outcomes: The spasticity in the neck will affect motor function of the whole body. There will be decreased stride length and arm swing on the side of the body with the neck muscle spasm. The shoulder girdle and pelvis will be continuously rotated around a vertical axis the same direction as the head in reference to the feet and direction of walking. The shoulder and pelvic girdles will be tilted such that they are closer together on one side than the other side due to side-bending of the torso. We also expect that there will be an indirect relationship between age and motor function. OMM is expected to significantly improve motor function and quality of life.

Significance: The impact of the neck muscle spasticity on full body biomechanics of subjects with primary cervical dystonia is not well understood, and the results can be used to improve assessment of function as well as management of the disorder.

Aim II. To determine whether osteopathic manual medicine used during the first four weeks following botulinum toxin intramuscular injection will significantly improve the joint range of motion, motor function, and quality of life of subjects with primary cervical dystonia .

Hypothesis II: Osteopathic manual medicine will improve the range of motion of the neck, symmetry of posture and gait, and quality of life of subjects with primary cervical dystonia.

Experimental approach: Subjects being treated with botulinum toxin injections will be evaluated with a standard spasmodic torticollis form (to be filled out by physician), cervical dystonia questionnaire regarding quality of life, and Vicon 3-Dimensional gait and posture analysis before and after four weekly treatments with OMM (n≥8) for comparison with subjects in a no-OMM control condition (n≥ 8).

Expected outcomes: Subjects will have improved quality of life in regard to head and neck symptoms, pain and discomfort, upper limb activities, walking, sleep, annoyance, mood, and psychosocial functioning. Subjects will have improved joint range of motion and motor function.

Significance: Although physicians specializing in osteopathic manual medicine treat patients with various types of dystonia, the effectiveness of osteopathic manual medicine in treating primary cervical dystonia is not established, and thus, osteopathic manual medicine is not recognized or recommended as adjunctive therapy. The botulinum toxin is injected into spastic neck muscles. However, there is no adjunctive procedure recommended for treating the rest of the symptoms associated with the illness. 3-dimensional characterization of motor function has been used in children with cerebral palsy and generalized dystonia before and after surgical intervention, and using a similar method may demonstrate how OMM can prevent people from becoming disabled.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cervical dystonia or spasmodic torticollis
* ages 2-100

Exclusion Criteria:

* no clinical diagnosis of cervical dystonia or spasmodic torticollis
* symptoms beginning over the age of 40
* pregnant women are excluded from Aim 2

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in Motor Function | baseline and 5 weeks
  Motor function will be assessed by Vicon 3-Dimensional analysis of the subjects' biomechanics while walking and will depict stride length and arm swing on each side of the body as well as the posture of the shoulder and pelvic girdle with reference to the coronal, transverse and sagittal planes.

SECONDARY OUTCOMES:
Change in Quality of Life | baseline and 5 weeks
  Quality of Life will be assessed by the CDIP-58 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jayme Mancini, DO, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided